CLINICAL TRIAL: NCT05496751
Title: Response Variability to Exercise in Adults
Brief Title: Response Variability to Exercise
Acronym: REVISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Ross, PhD (Other)
Responsible Party: Sponsor-Investigator, Robert Ross, PhD, Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ross2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Exercise; Cardiorespiratory Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low amount, low intensity exercise (Experimental): exercise dose (amount and intensity) will be controlled.
  Interventions: Behavioral: Low amount, low intensity exercise
- Low amount, high intensity exercise (Experimental): exercise dose (amount and intensity) will be controlled.
  Interventions: Behavioral: Low amount, high intensity exercise
- Control (No Intervention): no exercise intervention
- High amount, high intensity exercise (Experimental): exercise dose (amount and intensity) will be controlled.
  Interventions: Behavioral: High amount, high intensity exercise

INTERVENTIONS:
Behavioral: Low amount, low intensity exercise — Participants will exercise under supervision. Exercise dose will vary by amount and intensity
  Arms: Low amount, low intensity exercise
Behavioral: Low amount, high intensity exercise — Participants will exercise under supervision. Exercise dose will vary by amount and intensity
  Arms: Low amount, high intensity exercise
Behavioral: High amount, high intensity exercise — Participants will exercise under supervision. Exercise dose will vary by amount and intensity
  Arms: High amount, high intensity exercise

SUMMARY:
In this proposal, the investigators challenge the assumption that following the physical activity guidelines implies benefit for ALL adults, and that if benefit is not achieved in response to first line therapy, it will be by simply exercising more. Thus, for improving cardiorespiratory fitness and cardiometabolic risk factors, unanswered questions include: 1) To what extent, regardless of increasing exercise intensity or amount, is exercise not associated with benefit? Demonstration of a resistance to benefit through exercise in a substantial number of adults would be a novel and important finding, would counter the assumptions of many if not most health care practitioners, and could have immediate and direct application in all health care settings. 2) To what extent will non-responders to first line therapy (150 min/wk) be required to increase exercise intensity or amount to achieve benefit? 3) To what extent will failure to improve CRF segregate (be associate with) with cardiometabolic risk factors? The investigators propose that adults who remain exercise resistant for improvement in CRF and cardiometabolic risk despite increasing amount or intensity are at high risk of metabolic disease and consequently, are candidates for alternative treatment strategies.

DETAILED DESCRIPTION:
The trial has two objectives:

Primary objective: After 16 weeks of first line therapy (150 min/wk of MPA), does increasing exercise intensity or amount for 16 weeks improve cardiorespiratory fitness (CRF, VO2peak) deferentially depending on the CRF response at 16 weeks.

Secondary objective: Determine whether common cardiometabolic risk factors segregate/cluster with respect to variation in CRF to first line therapy in adults, and, whether clinically meaningful improvements in cardiometabolic risk factors segregate with improvement in CRF.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle (planned physical activity for one day per week or less).
* Weight stable (± 2 kg) for 6 months prior to the beginning of the study.
* BMI between 20 and 40 kg/m2.

Exclusion Criteria:

* Physical impairment which would make the intervention very difficult or unsafe according to doctor's advice.
* Diabetes, current smokers.
* Plan to move from the area in next 8 months.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | Measured at baseline and every 4 weeks for 32 weeks.
  Cardiorespiratory fitness will be determined using direct (open circuit spirometry) measures of oxygen consumption (expressed in L/min) obtained during a maximal treadmill test.

SECONDARY OUTCOMES:
Change in glucose | Measured at baseline, 16 and 32 weeks.
  Fasting glucose (mmol/L)
Change in blood lipids | Measured at baseline, 16 and 32 weeks.]
  Fasting LDL- and HDL-cholesterol (mmol/L)
Change in insulin | Measured at baseline, 16 and 32 weeks.]
  fasting insulin (pmol/L)
Change in triglycerides | Measured at baseline, 16 and 32 weeks.
  fasting triglycerides (mmol/L)
Change in body fat | Measured at baseline, 16 and 32 weeks
  Total adiposity
Change in abdominal fat | Measured at baseline, 16 and 32 weeks.
  Visceral adiposity
Change in lean body mass | Measured at baseline 16 and 32 weeks.
  Lean mass
Change in subcutaneous fat | Measured at baseline, 16 and 32 weeks.
  Subcutaneous adiposity
Change in obesity phenotype | Measured at baseline 16 and 32 weeks.
  waist circumference
Change on body weight | Measured at baseline, 16 and 32 weeks.
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Health Studies, Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All data will be made available upon request.
Time Frame: Within 1 year of study completion.
Access Criteria: Deidentified participant data collected during the trial will be available to external groups upon scientific review.

REFERENCES:
- [Derived] Ross R, Day AG, Stotz PJ, Wade S, Cooke R, Miller E, Liberatore N, Lamarche B. Response variability to exercise (REVISE): Study rationale, design and methods. Contemp Clin Trials Commun. 2025 Jul 5;46:101519. doi: 10.1016/j.conctc.2025.101519. eCollection 2025 Aug. PMID 40688055